CLINICAL TRIAL: NCT05262504
Title: Comparison of Visual Performance and Quality of Life With a Novel Non-diffractive Extended Depth-of-focus IOL and a Trifocal IOL
Brief Title: Comparison of a Novel Non-diffractive Extended Depth of Focus Intraocular Lens (IOL) and a Trifocal IOL
Status: Completed | Type: Observational
Sponsor: Baskent University Ankara Hospital (Other)
Responsible Party: Principal Investigator, Leyla Asena, Assoc. Prof. Dr., Baskent University Ankara Hospital
Other Study IDs: Vivity Panoptix
Record Dates: First submitted 2022-02-21; First posted 2022-03-02 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Intraocular Lens; Cataract; Quality of Life
Keywords: cataract; wavefront shaping; extended depth of focus; trifocal; intraocular lens; quality of life; defocus curve; contrast sensitivity; photic disturbance
MeSH Terms: conditions — Cataract | interventions — Lens Implantation, Intraocular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- EDOF IOL Group: Patients who were implanted with the novel wavefront shaping extended depth of focus IOL
  Interventions: Device: İntraocular lens implantation
- Multifocal IOL group: Patients who were implanted with the multifocal IOL
  Interventions: Device: İntraocular lens implantation

INTERVENTIONS:
Device: İntraocular lens implantation — Each participant underwent bilateral sequential cataract surgery and bilateral implantation of a novel non-diffractive EDOF IOL (n=26) or a trifocal IOL (n=26). The interval between the first and second-eye surgeries was 1 to 3 weeks. The patients selected the IOL model after they were fully informed regarding the advantages and disadvantages of each IOL, by their surgeon. Their degree of interest in greater spectacle freedom at far, intermediate, and near distances, as well as their daily activities such as frequency of night driving or reading habits were discussed. The possibility of photic disturbances was described and explained as well.

SUMMARY:
The purpose of this study is to compare visual performance and quality of life (QOL) following bilateral implantation of a novel non-diffractive extended depth-of-focus (EDOF) intraocular lens (IOL) (AcrySof® IQ Vivity, Alcon, TX, USA) and a trifocal IOL (Acrysof® IQ PanOptix, Alcon, Fort Worth, TX) in a prospective comparative interventional case series.

DETAILED DESCRIPTION:
Developments in cataract surgical devices and intraocular lenses (IOL) increased patient expectations and changed the practice patterns in ophthalmology. Nowadays, cataract surgery is considered as a refractive surgery. With multifocal IOLs, spectacle independence can be achieved with a good distance, intermediate and near visual acuity. This is associated with increased quality of life after cataract surgery.The most important disadvantages of multifocal IOLs are loss of contrast sensitivity and photic phenomena such as glare and halo. Although multifocal IOLs are more frequently associated with photic disturbances than monofocal IOLs, the trifocal IOLs have improved performance in photic phenomena when compared to bifocal IOLs. Recently, a new technology known as extended depth of focus (EDOF) IOLs have been developed. These lenses create a single elongated focal point to enhance the depth of focus, improving intermediate vision without compromising distance vision. Although EDOF IOLs provide better intermediate distance vision when compared to monofocal IOLs, near vision is not as good as trifocal IOLs. The most important advantage provided by the EDOF technology is lower rate of photic disturbances than trifocal IOL designs. The aim of this study was to compare the visual performance and patient-reported quality of life (QOL) outcomes following bilateral implantation of a novel non-diffractive wavefront shaping EDOF IOL (AcrySof® IQ Vivity, Alcon Research, TX, USA) and a trifocal IOL (AcrySof® IQ PanOptix, Alcon Laboratories, Fort Worth, TX).

ELIGIBILITY:
Inclusion Criteria:

* Cataract patients scheduled for surgery who are interested in spectacle independence.
* Bilateral cataract with plan of bilateral sequential cataract surgery.
* Adult patients older than 18 years of age
* Normal cognitive function, able to understand advantages and disadvantages associated with different types of IOLs.

Exclusion Criteria:

* Ocular diseases other than cataract including irregular astigmatism, diabetic retinopathy, age-related macular degeneration or any other retinal diseases, severe dry eye, glaucoma, amblyopia, uveitis, pseudoexfoliation syndrome, abnormal pupillary function, history of intraocular or corneal surgery, congenital eye abnormalities, or eye trauma.
* Patients with high myopia with axial length (AL) ≥ 26,5 mm and high hyperopia (AL ≤ 21.5 mm)
* Lifestyle and work-related factors requiring sharp near or distance vision
* Patients with unrealistic visual expectations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 104 eyes of 52 consecutive patients with bilateral cataracts operated between April and September 2021 were included. All patients were interested in spectacle independence. Each participant underwent bilateral sequential cataract surgery and bilateral implantation of a novel non-diffractive EDOF IOL (n=26) or a trifocal IOL (n=26). The patients selected the IOL model after they were fully informed regarding the advantages and disadvantages of each IOL, by their surgeon. Their degree of interest in greater spectacle freedom at far, intermediate, and near distances, as well as their daily activities such as frequency of night driving or reading habits were discussed. The possibility of photic disturbances was described and explained as well.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Postoperative visual acuity with or without spectacle correction at near, far and intermediate distances | postoperative third month
  uncorrected distance visual acuity (UDVA), corrected distance visual acuity (CDVA), distance corrected intermediate visual acuity (DCIVA), distance corrected near visual acuity (DCNVA)
Defocus-curves | postoperative third month
  The monocular defocus curves were evaluated under photopic conditions using defocusing lenses from +0.50 D to -4.00 D in 0.50 D steps. The measurements were performed by adding the lenses to the CDVA.
Contrast sensitivity | postoperative third month
  Monocular and binocular contrast sensitivity was assessed with the Pelli-Robson chart under photopic conditions at 3 meters.
Reading speed | postoperative third month
  Reading speed was measured using the validated Turkish version of the MNREAD chart in photopic illumination conditions. It was recorded as number of words read by the patient in one minute (words per minute-wpm).
Quality of vision / dysphotopsia | postoperative third month
  Dysphotopsia was assessed by the Quality of Vision (QoV) questionnaire developed by McAlinden et al. The QoV is a validated Rasch-adjusted questionnaire in which patients are asked to rate specific dysphotopsia items depicted in standard photographs. Patients score each item (0, 1, 2, or 3) in relation to how frequent, severe, and bothersome their symptoms are (30 items in total). Lower QoV scores indicate a better quality of vision.
Vision-related quality of life (QOL) | postoperative third month
  The vision-related QOL was assessed three months after the surgery by the VF-14 QOL questionnaire that was administered face-to-face by a trained researcher (İK). The grading scale was as follows: 0, no difficulty; 1, a little difficulty; 2, moderate difficulty; 3, quite difficult; 4, impossible to perform. Special care was taken not to influence the patients and to ensure that each question was fully understood.

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Oto, MD, Study Chair — Baskent University Faculty of Medicine Department of Ophthalmology
Locations (1):
- Baskent University Faculty of Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Data will be available upon request.

REFERENCES:
- [Derived] Asena L, Kirci Dogan I, Oto S, Dursun Altinors D. Comparison of visual performance and quality of life with a new nondiffractive EDOF intraocular lens and a trifocal intraocular lens. J Cataract Refract Surg. 2023 May 1;49(5):504-511. doi: 10.1097/j.jcrs.0000000000001142. PMID 36700928